CLINICAL TRIAL: NCT03450265
Title: A Randomized, Controlled, Non-inferiority Study to Evaluate the Efficacy and Safety of Hemopatch Compared to TachoSil in Preventing or Reducing Postoperative Air Leaks After Pulmonary Resection
Brief Title: Hemopatch Compared to TachoSil in Postoperative Air Leak Duration After Pulmonary Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BXU513667; 2017-003931-12 (EudraCT Number)
Record Dates: First submitted 2018-02-13; First posted 2018-03-01 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Air Leak From Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemopatch (Experimental): Patients undergo elective pulmonary resection. Following resection, primary stapling and suturing will be done and air leakage will be assessed. If a specific grade-level of air leakage is present, patients will be randomized and either Hemopatch or TachoSil applied.
  Interventions: Device: Hemopatch
- TachoSil (Active Comparator): Patients undergo elective pulmonary resection. Following resection, primary stapling and suturing will be done and air leakage will be assessed. If a specific grade-level of air leakage is present, patients will be randomized and either Hemopatch or TachoSil applied.
  Interventions: Device: Tachosil

INTERVENTIONS:
Device: Hemopatch — Applied according to the current instruction for use (IFU). According to the IFU, a maximum of 7 Hemopatch 45 x 90 mm patches can be used in adults.
  Arms: Hemopatch
Device: Tachosil — Applied according to the current instruction for use (IFU).
  Arms: TachoSil

SUMMARY:
This study is a randomized, controlled study, with the primary objective to demonstrate non-inferiority of Hemopatch compared to TachoSil in postoperative air leak duration after pulmonary resection, and with the secondary objective of evaluating the safety of Hemopatch compared to TachoSil.

ELIGIBILITY:
Inclusion Criteria:

Preoperative-

* Patients, 18 years or older at the time of signing the informed consent form (ICF), undergoing elective pulmonary resections (lobectomy, segmentectomy, or wedge resection), either through open thoracotomy or through Visually Assisted Thoracotomy surgery (VATS)
* Patients or legally authorized representatives, who are able to give IC after an explanation of the proposed study, and who are willing to comply with the study requirements for therapy during the entire study treatment period
* If female of child-bearing potential, patient will present with a negative blood/urine pregnancy test, and will agree to employ adequate birth control measures for the duration of the study

Intraoperative-

* Patients with grade 1 or 2 (Macchiarini scale) air leakage after primary stapling and limited suturing

Exclusion Criteria:

Preoperative-

* Patients who had previous lung surgery (on the same side)
* Patients with an active, florid infection
* Patients who have received chemotherapy within the previous 3 weeks.
* Patients who have received radiation therapy within the previous 4 weeks.
* Patients with known hypersensitivity to the components of the investigational product and control (human fibrinogen, human thrombin, collagen of any origin, NHS-PEG)
* Patients undergoing emergency surgery
* Female patients of childbearing potential with a positive pregnancy test or intent to become pregnant during the clinical study period
* Female patients who are nursing
* Patients with exposure to another investigational drug or device clinical trial within 30 days prior to enrollment or anticipated in the 30 day study period till the End of study visit.
* Patient has a clinically significant concurrent medical condition (e.g. concomitant illness, drug/alcohol abuse) that, in the opinion of the investigator, could adversely affect patient's safety and/or compliance with study procedures
* Patient is a family member or employee of the investigator

Intraoperative-

* Patients with serious complications during surgery, including the need for adhesiolysis, and pneumonectomy.
* Patients who were treated with any surgical sealant
* Major intraoperative complications that require resuscitation or deviation from the planned surgical procedure
* Patients with any other intraoperative findings identified by the surgeon that may preclude the conduct of the study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative air leakage | Day 1 to Day 30

SECONDARY OUTCOMES:
Incidence of intraoperative treatment failure | Day 1
Incidence of patients with prolonged air leakage defined as air leakage > 5 Days | Day 5 to Day 30
Number of additional procedures needed | Day 1 to Day 30
  Type of procedures include chest drainage, re-operation, respiratory assistance, and blood transfusion
Time to chest tube removal | Day 1 to Day 30
Time in surgery (minutes) from incision to closure | Day 1
Length of stay in hospital (days) | Day 1 to Day 30
Number of unplanned interventions | Day 1 to Day 30
Incidence of pre-defined postoperative Adverse Events of Special Interest (AESIs) | Day 1 to Day 30
  Pre-defined AEs include Pneumothorax, Bronchopleural fistula, Emphysema (subcutaneous and mediastinal), Pleural effusions, Postoperative respiratory failure, Empyema, Allergic reactions in reasonable temporal relationship with the product application
Number of patches used intra-operatively | Day 1

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (5):
  - Baxter Investigational Site, Catania
  - Baxter Investigational Site, Milan
  - Baxter Investigational Site, Padua
  - Baxter Investigational Site, Pisa
  - Baxter Investigational Site, Rome
- Spain (5):
  - Baxter Investigational Site, Seville, Andalusia
  - Baxter Investigational Site, Madrid, Getafe
  - Baxter Investigational Site, Madrid, Madrid
  - Baxter Investigational Site, Alzira, Valencia
  - Baxter Investigational Site, Madrid